CLINICAL TRIAL: NCT03812991
Title: The Use of Intranasal Calcitonin to Improve Pain and Activity in Elderly Pelvic Ring Injuries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett D. Crist, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013172
Record Dates: First submitted 2019-01-11; First posted 2019-01-23 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pelvic Ring Fractures
MeSH Terms: interventions — salmon calcitonin; Calcitonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Non-Treatment Group (No Intervention): This is the Non-Treatment Arm of the study. No intervention is to be administered.
- Miacalcin Calcitonin Salmon Nasal Spray (Experimental): 1 spray (200 IU) qDay, alternate nostrils daily
  Interventions: Drug: Miacalcin Calcitonin Salmon Nasal Spray

INTERVENTIONS:
Drug: Miacalcin Calcitonin Salmon Nasal Spray — Miacalcin nasal spray is 1 spray (200 International Units) per day administered intranasally, alternating nostrils daily
  Other Names: Miacalcin; Calcitonin
  Arms: Miacalcin Calcitonin Salmon Nasal Spray

SUMMARY:
Pelvic ring fractures in the geriatric population are a rising problem for surgeons in industrialized countries. Many of these low-energy fractures are treated nonoperatively; however, pain is a significant factor in recovery of these patients and often inhibits their ability to mobilize. Most of these fractures are lateral compression type 1 injuries which are defined as an impaction to the sacrum with varying amounts of anterior/pubic root/rami fractures. Many of these patients in the geriatric population suffer from osteoporosis and the injuries are often sustained from a low-energy mechanism like a fall. The tenet of treatment for all osteoporotic fractures is early mobilization. It is well known that extended periods of bed rest will lead to pneumonia, decubitus ulceration, deep venous thrombosis, and, in the case of the pelvis, not prevent subsequent deformity. Calcitonin is a polypeptide containing 32 amino acids, and it plays a role in the regulation of bone metabolism as a hormone that prevents bone resorption. Intranasal salmon calcitonin (ISC) has been demonstrated to decrease pain and improve the level of activity in patients with acute vertebral osteoporotic compression fractures when administered within the first 5 days of onset of pain/injury. It has also demonstrated an immediate post analgesic effect in osteoporotic distal radius fractures treated nonoperatively. The antihyperalgesic action of calcitonin appears to be mediated by serotonin receptors. The purpose of this study is to evaluate the analgesic effect of ISC on geriatric patients with pelvic ring injuries who are treated nonoperatively.

DETAILED DESCRIPTION:
Baseline: Treatment group will be prescribed 200IU of ISC daily for a period of 3 months. The control group will not be prescribed calcitonin. Participants will complete research only Iowa pelvis score questionnaire, SF-36 questionnaire and visual analogue scale (VAS) to assess subjective pain and function. Two-week follow up visit post discharge: participants will complete Iowa pelvis score questionnaire, SF-36 questionnaire and VAS to assess subjective pain and function. Participants will be referred for a standard of care DEXA bone density scan if they have no previous diagnosis of osteoporosis and no history of previous scan within a year. Six weeks post discharge: participants will complete Iowa pelvis score questionnaire, SF-36 questionnaire and VAS to assess subjective pain and function. Participants will undergo standard of care radiographic analysis of pelvic ring injury with AP/inlet and outlet pelvic x-rays 4. Twelve weeks post discharge: Participants will complete Iowa pelvis score questionnaire, SF-36 questionnaire and VAS to assess subjective pain and function. Participants will undergo standard of care radiographic analysis of pelvic ring injury with AP/inlet and outlet pelvic x-rays - Participants will perform a timed up and go (TUG) test.

After informed consent is obtained, all patients who meet eligibility criteria will be randomized into one of two groups. Randomization will be achieved by numbering 50 sealed white envelopes (25 control, 25 treatment). There is no blinding to the randomization. It would be difficult to blind the participants, or the research personnel. We do not believe there will be any significant bias that can be corrected with blinding.

Treatment: 200IUof ISC daily for a period of 3 month

Control: Will not be prescribed calcitonin (ISC)

ELIGIBILITY:
Inclusion Criteria:

•Males or females over the age of 65 who sustain isolated pelvic ring injuries via a low-energy mechanism

Exclusion Criteria:

* An open pelvic ring fracture
* Concomitant acetabular fracture
* They are on ISC prior to enrollment
* Allergic or have contraindications to calcitonin or salmon
* Sustain other injuries in their spine or lower extremities
* Unwilling to participate in the study
* Nonambulatory at baseline
* Neurologic deficit associated with the pelvic ring injury

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health System, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Treatment Group | Miacalcin Calcitonin Salmon Nasal Spray
Started | 11 | 10
Completed | 8 | 9
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Population: Only participants who completed the study are included in the analysis of the data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Treatment Group | Miacalcin Calcitonin Salmon Nasal Spray | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Full Range); unit: Years] | 81 [65 to 95] | 81 [65 to 93] | 81 [65 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale
Description: Compare acute pain using (Visual Analogue Scale on a scale of 0-10 with 0=no pain and 10= worst pain imaginable.
Time Frame: The subject will be enrolled/assessed up to three months post-injury.
Population: Only participants who completed the study are included in the analysis of the data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Treatment Group | Miacalcin Calcitonin Salmon Nasal Spray
Number analyzed (Participants) | 8 | 9
units on a scale
  Baseline | 6.0 (2.0) | 6.8 (2.8)
  2 Week Follow Up | 5.5 (2.2) | 3.7 (3.0)
  6 Week Follow Up | 5.2 (3.0) | 2.0 (2.3)
  3 Month Follow Up | 1.9 (1.4) | 2.2 (2.3)

2. Secondary Outcome: Iowa Pelvic Score (IPS)
Description: IPS is a questionnaire with 6 items subsets which are totalled to assess functional outcomes in pelvic ring injury patients. The total will range from 15 - 100 with a higher total score being associated with a better outcome.
  1. activities of daily life (20 activities of daily living asking if participant can perform requiring a Yes / No response) with Yes =1, No =0. Subset Min= 0 Max=20.
  2. work history (no change = 20, Fulltime, change =15, Part-Time=10, Unable=5) Subset Min= 5 Max = 20.
  3. pain (None, not significant=25, Occasional medication=20, Regular medication=15, Hospitalization/operation=5) Min = 5 Max= 25.
  4. limping (None=20, Yes=15, Appliance=10), and Non-ambulatory=5) Min=5 Max=20.
  5. visual pain line (visual analogue scale) (Scale of 0-10 with 0=no pain and 10=worst imaginable pain) Min=0 Max=10 with higher score associated with a worse outcome.
  6. cosmesis (No significance=5 and Significant change=0).
Time Frame: The subject will be enrolled/assessed up to three months post-injury.
Population: Only participants who completed the study are included in the analysis of the data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Treatment Group | Miacalcin Calcitonin Salmon Nasal Spray
Number analyzed (Participants) | 8 | 9
score on a scale
  Baseline | 70.5 (18.0) | 64.5 (12.0)
  2 Weeks Follow Up | 57.2 (27.0) | 47.3 (10.0)
  6 Weeks Follow Up | 65.7 (10.0) | 66.3 (12.0)
  3 Month Follow Up | 71.0 (11.0) | 71.5 (9.0)

3. Secondary Outcome: SF-36 Short Form Health Survey
Description: SF-36 Short Form Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Note that all items are scored so that a high score defines a more favorable health state.
  Each item in a scale is scored on a 0-100 range, each scale is averaged to create 8 scale scores. These scores are linearly transformed onto a scale from 0 (negative health) to 100 (positive health).
Time Frame: The subject will be enrolled/assessed up to three months post-injury.
Population: Only participants who completed the study are included in the analysis of the data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Treatment Group | Miacalcin Calcitonin Salmon Nasal Spray
Number analyzed (Participants) | 8 | 9
score on a scale
  Baseline | 59.4 (33.0) | 56.3 (9.0)
  2 Week Follow Up | 58.8 (18.0) | 52.7 (16.)
  6 Week Follow Up | 59.6 (13.0) | 53.8 (12.0)
  3 Month Follow Up | 58.8 (18.0) | 53.8 (12.0)

4. Secondary Outcome: Timed Get Up and Go (TUG)
Description: The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down with scoring as noted:
  < 10 seconds = normal < 20 seconds = good mobility; can walk outside alone; does not require a walking aid < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid
Time Frame: The subject will be assessed at the three months post-injury
Population: Only participants who completed the study are included in the analysis of the data.
Measure: Mean (Standard Deviation); unit: "seconds"
Arm/Group | Non-Treatment Group | Miacalcin Calcitonin Salmon Nasal Spray
Number analyzed (Participants) | 8 | 9
"seconds" | 13.7 (5.5) | 13.3 (3.0)

5. Secondary Outcome: Radiographic Healing Using Intranasal Salmon Calcitonin
Description: To compare radiographic healing using AP/inlet and outlet pelvic x-rays on geriatric patients with pelvic ring injuries who receive intranasal salmon calcitonin and with those who do not receive intranasal salmon calcitonin.
Time Frame: Fracture healing and alignment will be assessed at six weeks and three months post-injury.
Population: Only participants who completed the study are included in the analysis of the data.
Measure: Number; unit: participants
Arm/Group | Non-Treatment Group | Miacalcin Calcitonin Salmon Nasal Spray
Number analyzed (Participants) | 8 | 9
participants
  6 Week Follow Up | 8 | 9
  3 Month Follow Up | 8 | 9

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and other nonserious adverse events were not assessed for study participants in this study.
Arm/Group | Non-Treatment Group | Miacalcin Calcitonin Salmon Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03812991/Prot_001.pdf